CLINICAL TRIAL: NCT03051893
Title: A Two-part Open Label, Randomised, Single Dose, Crossover Study in Healthy Volunteers to: (Part A) Compare the Pharmacokinetics of up to 6 Chronocort® Formulations, and (Part B) Determine the Dose Proportionality of a Selected Chronocort® Formulation at Three Dose Levels With an Additional Comparison With the Selected Formulation Dosed on Two Occasions Over a 24 Hour Period
Brief Title: A Two-part, Study to Compare the Pharmacokinetics and Dose Proportionality of up to 6 Chronocort Formulations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Neurocrine UK Limited (Industry)
Collaborators: Simbec Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DIUR-002
Record Dates: First submitted 2017-01-11; First posted 2017-02-14 (Actual); Last update posted 2017-02-14 (Actual); Status verified 2017-02

CONDITIONS: Adrenal Insufficiency; Congenital Adrenal Hyperplasia
MeSH Terms: conditions — Adrenal Insufficiency; Adrenal Hyperplasia, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Part A1 (Experimental): Three formulations of Chronocort 30mg were administered to healthy volunteers, with a 7-day washout period between each dose. Each treatment was administered in a randomised, crossover manner.
  Interventions: Drug: Chronocort
- Part A2 (Experimental): Three additional formulations of Chronocort 30mg were administered to healthy volunteers, with a 7-day washout period between each dose. Each treatment was administered in a randomised, crossover manner.
  Interventions: Drug: Chronocort
- Part B (Experimental): The best formulation of Chronocort was then selected from Parts A1 & A2. This was then administered in four separate treatment periods, in dosages of 5mg, 10mg, 20mg and 30mg. Each treatment was administered in a randomised, crossover manner.
  Interventions: Drug: Chronocort

INTERVENTIONS:
Drug: Chronocort — Modified formulation of hydrocortisone

SUMMARY:
This was an open label, randomised, single dose study, comprising Part A (undertaken in two separate three-period crossover cohorts denoted as A1 and A2) and Part B (undertaken in one four-period crossover cohort), to evaluate the PK of Chronocort® in healthy male volunteers. The washout interval in both Part A and Part B was 1-week in between each treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers between 18 and 60 years of age, inclusive (at screening).
* Subjects with a Body Mass Index (BMI) of 21-28. Body Mass Index = Body weight (kg) / (Height (m))2.
* Subjects with no clinically significant abnormal serum biochemistry, haematology and urine examination values within 14 days prior to the first dose.
* Subjects with negative urinary drugs of abuse screen determined within 14 days prior to the first dose.
* Subjects with negative HIV and Hepatitis B and C results.
* Subjects with no clinically significant abnormalities in 12-lead electrocardiogram (ECG) determined within 14 days prior to the first dose.
* Subjects with no clinically-significant deviation outside the normal ranges for blood pressure and pulse measurements.
* Subjects and sexual partners used effective contraception methods during the trial and for 3 months after the last dose, for example:

  * Oral contraceptive and condom
  * Intra-uterine device (IUD) and condom
  * Diaphragm with spermicide and condom
* Subjects were available to complete the study.
* Subjects satisfied a medical examiner about their fitness to participate in the study.
* Subjects provided written informed consent to participate in the study.
* Subject continued to meet all screening inclusion criteria prior to dosing.
* Subjects with no clinically significant abnormal serum biochemistry, haematology and urine examination values including negative urinary drugs of abuse screen (including alcohol) prior to dosing.

Exclusion Criteria:

* A clinically significant history of gastrointestinal disorder likely to influence drug absorption.
* Receipt of regular medication within 14 days prior to the first dose (including high dose vitamins, dietary supplements or herbal remedies).
* Receipt of any vaccination within 14 days prior to the first dose.
* Evidence of renal, hepatic, central nervous system, respiratory, cardiovascular or metabolic dysfunction.
* Presence of clinically significant infections (systemic fungal and viral infections, acute bacterial infections)
* Current or previous history of tuberculosis
* A clinically significant history of previous allergy / sensitivity to Hydrocortisone and/or Dexamethasone.
* A clinically significant history or family history of psychiatric disorders/illnesses.
* A clinically significant history of drug or alcohol abuse.
* Inability to communicate well with the Investigator (i.e., language problem, poor mental development or impaired cerebral function).
* Participation in a New Chemical Entity clinical study within the previous 16 weeks or a marketed drug clinical study within the previous 12 weeks. (N.B. The washout period between trials was defined as the period of time elapsed between the last dose of the previous study and the first dose of the next study)
* Subjects who have consumed more than 2 units of alcohol per day within seven (7) days prior to the first dose or have consumed any alcohol within the 48 hour period prior to the first dose.
* Donation of 450ml or more of blood within the previous 12 weeks.
* Subjects who smoked (or ex-smokers who had smoked within 6 months prior to first dose).
* Subjects who worked shifts (i.e. regularly alternated between days, afternoons and nights).

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2011-02; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
To compare the Tmax of six formulations of Chronocort® (30 mg, dosed at night) over an 18 hour period. Parts A1 & A2 only | 18 hours
  Time at maximum concentration in serum
To compare the Cmax of six formulations of Chronocort® (30 mg, dosed at night) over an 18 hour period. Parts A1 & A2 only | 18 hours
  Maximum serum concentration
To compare the AUC0-t of six formulations of Chronocort® (30 mg, dosed at night) over an 18 hour period. | 18 hours
  Area under the plasma concentration-time curve
To compare the AUC0-∞ of six formulations of Chronocort® (30 mg, dosed at night) over an 18 hour period. | 18 hours
  Area under the plasma concentration-time curve from zero (0) hours to infinity (∞)
To compare the CL of six formulations of Chronocort® (30 mg, dosed at night) over an 18 hour period. | 18 hours
  Drug clearance (CL) is defined as the volume of plasma in the vascular compartment cleared of drug per unit time

CONTACTS AND LOCATIONS:
Overall Officials: Girish Sharma, Principal Investigator — Simbec Research

IPD SHARING:
Plan to Share IPD: No